CLINICAL TRIAL: NCT06536595
Title: Validity and Reliability of the Turkish Version of the Hand Scleroderma Lived Experience Scale
Brief Title: Validity and Reliability of the Turkish Version of HAnDE
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gamze Pala, Research assistant, Gazi University
Other Study IDs: 2021-1
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Scleroderma; Hand Rheumatism
Keywords: hand; reliability; scale; validation; scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: got diagnosed scleroderma
  Interventions: Other: Scales

INTERVENTIONS:
Other: Scales — Participants were asked to complete the HAnDE-T, MHISS, SF-36 and HAQ when they first came. After 1 week, they were asked to complete HAnDE-T for re-test.

SUMMARY:
The aim of the present study was to translate and cross-culturally adapt The Hand Scleroderma Experienced Experience (HAnDE) Scale into the Turkish language and investigate its reliability and validity in Turkish-speaking patients with systemic sclerosis.

DETAILED DESCRIPTION:
Objective: The aim of the present study was to translate and cross-culturally adapt The Hand Scleroderma Experienced Experience (HAnDE) Scale into the Turkish language and investigate its reliability and validity in Turkish-speaking patients with systemic sclerosis.

Methods: The HAnDE was cross-culturally adapted according to Beaton's guideline. Participants completed the Turkish version of HAnDE scale (HAnDE-T), The Mouth Handicap in Systemic Sclerosis Scale (MHISS), 36 Item Short Form Survey (SF-36), Health Assessment Questionnaire (HAQ). Internal consistency of the HAnDE-T questionnaire was evaluated by Cronbach's alpha coefficient. Convergent validity was tested using Pearson's correlation coefficient. The construct validity of the HAnDE-T questionnaire was assessed by factor analysis. The construct validity of the HAnDE-T was evaluated by correlating the scores between HAnDE-T and HAQ, SF-36 PCS, SF-36 MCS and MHISS scores.

ELIGIBILITY:
Inclusion Criteria:

* 1) being 18-65 years of age,
* 2) being diagnosed of SSc according to do 2013 American College of Rheumatology (ACR) criteria and/or European League Against Rheumatism (EULAR) criteria,
* 3) being literate in Turkish,
* 4) being agreed to participate in the research.

Exclusion Criteria:

* 1) being in a psychological or cognitive disorders that would prevent to answer questions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diagnosed with scleroderma
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
HAnDE-T | Patients were asked to complete the HAnDE-T when they first came (baseline). After 1 week, they were asked to complete HAnDE-T for retest.
  The Hand Scleroderma Lived Experience Scale. HAnDE is a PROM scale developed by Sibeoni et al. to assess the patient's current situation regarding his/her lived experience of global hand involvement. It consists of 16 questions that patients answer by giving a score between 0 and 4. While 0 means "I do not agree at all", 4 means "I completely agree." The total score of the HAnDE is determined by the sum of all answers given. The total score ranges from 0 to 64. Higher scores indicated higher hand involvement.

SECONDARY OUTCOMES:
MHISS | Patients were asked to complete the MHISS when they first came (baseline).
  The Mouth Handicap in Systemic Sclerosis Scale. MHISS is a scale developed by Mouthon et al. to quantify the handicap associated with mouth disability in patients with SSc. The MHISS consists of 12 questions to assess mouth-related disability. Patients responded to each question by giving a score of at least 0 and maximum 4. MHISS includes three domains: mouth opening, mouth dryness and esthetic concerns. The score that can be obtained from the scale ranges from 0 to 48, with higher scores indicating more limitations. The Turkish version of the MHISS was shown to be valid and reliable.
SF-36 | Patients were asked to complete the SF-36 when they first came (baseline).
  36-Item Short Form Survey. The SF-36 is a general quality of life assessment scale widely used to assess the quality of life. It was developed by the Rand Corporation in 1992. The SF-36 is a scale consisting of 8 sections and 36 items, including physical functionality, role limitations due to physical health problems, pain, social functionality, general health status, role limitations due to emotional problems, energy/vitality and mental health. The scale gives the total score for each subscale separately. The total score ranges from 0 to100. 0 indicates "poor health" status, 100 indicates "good health" status. The Turkish version of the SF-36 was shown to be valid and reliable.
HAQ | Patients were asked to complete the HAQ when they first came (baseline).
  Health Assessment Questionnaire. HAQ is an instrument developed to evaluate physical disability in 8 domains of the function: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activity. HAQ has been validated in patients with scleroderma. HAQ has 20 items in which patients evaluate their daily living activities by scoring between 0 and 3. The score of the test is determined by dividing the total scores given by the number of questions and varies between 0 and 3. The Turkish version of the HAQ was shown to be valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Deran Oskay, Prof. Dr., Study Director — Gazi University
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No